CLINICAL TRIAL: NCT03159416
Title: A Single-Dose, Open-Label, Parallel-Group Study to Assess the Pharmacokinetics of Inclisiran in Subjects With Renal Impairment Compared to Subjects With Normal Renal Function (ORION-7)
Brief Title: A Study of Inclisiran in Participants With Renal Impairment Compared to Participants With Normal Renal Function (ORION-7)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDCO-PCS-16-03
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — ALN-PCS

STUDY DESIGN:
Masking Description: Open-Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Inclisiran (normal renal function) (Experimental): Participants will receive a single dose of 300 milligram (mg) inclisiran administered by SC injection on Day 1. Normal renal function is defined as estimated creatinine clearance (CrCl) of ≥90 milliliter (mL)/minute (min).
  Interventions: Drug: Inclisiran
- Inclisiran (mild renal impairment) (Experimental): Participants will receive a single dose of 300 mg inclisiran administered by SC injection on Day 1. Mild renal impairment is defined as CrCl ranging from 60 to 89 mL/min.
  Interventions: Drug: Inclisiran
- Inclisiran (moderate renal impairment) (Experimental): Participants will receive a single dose of 300 mg inclisiran administered by SC injection on Day 1. Moderate renal impairment is defined as CrCl ranging from 30 to 59 mL/min.
  Interventions: Drug: Inclisiran
- Inclisiran (severe renal impairment) (Experimental): Participants will receive a single dose of 300 mg inclisiran administered by SC injection on Day 1. Severe renal impairment is defined as CrCl ranging from 15 to 29 mL/min.
  Interventions: Drug: Inclisiran

INTERVENTIONS:
Drug: Inclisiran — Inclisiran is a synthetic, chemically modified small interfering ribonucleic acid (siRNA) targeting proprotein convertase subtilisin kexin type 9 (PCSK9) messenger ribonucleic acid (mRNA) with a covalently attached triantennary N-acetylgalactosamine (GalNAc) ligand.
  Other Names: ALN-PCSSC

SUMMARY:
This study is a Phase I, single-dose, open-label trial to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics of a single dose of inclisiran subcutaneous (SC) injection in participants with mild, moderate, and severe renal impairment compared to participants with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants 18 to 80 years of age
* Participants should be qualified for inclusion based upon estimated CrCl ranges for normal renal function group and mild, moderate, and severe renal impairment groups

Exclusion Criteria:

* Participants with acute renal disease and/or history of renal transplant
* Urinary incontinence without catheterization
* Participants requiring hemodialysis
* Participants with LDL-C <60 mg/deciliter (dL) (or less than 1.55 millimoles/liter [mmol/L])
* Participants with Amyloid Kidney (if known by pathology)
* Participants with any significant hepatic, cardiac, or pulmonary disease or participants who are clinically nephritic

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2018-03-24 (Actual); Study Completion 2018-03-24 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Maximum Observed Plasma Concentration (Cmax) Of Inclisiran | 0 (pre-dose), 0.5, 1, 2, 4, 6, 8, 12, 24, and 48 hours post-dose and Day 4, Day 7, Day 14, and Day 30 post-dose
  Measurement of effect of renal impairment on PK of inclisiran by assessment of Cmax. Serial blood samples will be collected for the analysis. PK parameters will be determined from the plasma concentration-time profiles using a noncompartmental approach.
Pharmacokinetics: Tmax And t1/2 Of Inclisiran | 0 (pre-dose), 0.5, 1, 2, 4, 6, 8, 12, 24, and 48 hours post-dose and Day 4, Day 7, Day 14, and Day 30 post dose
  Measurement of effect of renal impairment on PK of inclisiran by assessment of time to reach maximum plasma concentration (Tmax) and time for inclisiran to reach half of its initial value (t1/2). Serial blood samples will be collected for the analysis. PK parameters will be determined from the plasma concentration-time profiles using a noncompartmental approach.
Pharmacokinetics: AUC0-24, AUC0-48, And AUC0-inf Of Inclisiran | 0 (pre-dose), 0.5, 1, 2, 4, 6, 8, 12, 24, and 48 hours post-dose and Day 4, Day 7, Day 14, and Day 30 post dose
  Measurement of effect of renal impairment on PK of inclisiran by assessment of area under the curve of the plasma concentration (AUC) from time 0 to 24 hours (AUC0-24), from time 0 to 48 hours (AUC0-48), and from time 0 extrapolated to infinity (AUC0-inf). Serial blood samples will be collected for the analysis. PK parameters will be determined from the plasma concentration-time profiles using a noncompartmental approach.
Pharmacokinetics: Apparent Total Clearance (CL/F) Following SC Administration Of Inclisiran | 0 (pre-dose), 0.5, 1, 2, 4, 6, 8, 12, 24, and 48 hours post-dose and Day 4, Day 7, Day 14, and Day 30 post dose
  Measurement of effect of renal impairment on PK of inclisiran by assessment of CL/F. Serial blood samples will be collected for the analysis. PK parameters will be determined from the plasma concentration-time profiles using a noncompartmental approach.
Pharmacokinetics: Vd/F During The Terminal Elimination Phase Following SC Administration Of Inclisiran | 0 (pre-dose), 0.5, 1, 2, 4, 6, 8, 12, 24, and 48 hours post-dose and Day 4, Day 7, Day 14, and Day 30 post dose
  Measurement of effect of renal impairment on PK of inclisiran by assessment of apparent volume of distribution (Vd/F) of inclisiran during the terminal elimination phase. Serial blood samples will be collected for the analysis. PK parameters will be determined from the plasma concentration-time profiles using a noncompartmental approach.
Pharmacokinetics: Amount Excreted Unchanged In Urine (Ae) Of Inclisiran Over 48 Hours Post-Dose | 0 up to 6 hours, 6 up to 12 hours, 12 up to 24 hours, and 24 up to 48 hour post-dose intervals
  Measurement of effect of renal impairment on PK of inclisiran by assessment of Ae of inclisiran. Pooled urine samples will be used for the analysis.
Pharmacokinetics: Fraction Excreted (Fe) Of Inclisiran | 0 up to 6 hours, 6 up to 12 hours, 12 up to 24 hours, and 24 up to 48 hour post-dose intervals
  Measurement of effect of renal impairment on PK of inclisiran by assessment of the urinary recovery rate over a specific collection interval (Fe), calculated as 100*Ae/Dose. Pooled urine samples will be used for the analysis.
Pharmacokinetics: Renal Clearance (CLr) Of Inclisiran | 0 up to 6 hours, 6 up to 12 hours, 12 up to 24 hours, and 24 up to 48 hour post-dose intervals
  Measurement of effect of renal impairment on PK of inclisiran by assessment of CLr, calculated as Ae/AUC0-48 plasma. CLr will be calculated if possible (for example, if the percent of unchanged drug excreted in urine exceeds 20%). Pooled urine samples will be used for the analysis.

SECONDARY OUTCOMES:
Change From Baseline In Lipids And Lipoproteins At Day 60 | Baseline, Day 60
  Pharmacodynamic effects of inclisiran on lipids and lipoproteins (total cholesterol, triglycerides, and high-density lipoprotein cholesterol, calculated and measured by beta-quant low-density lipoprotein cholesterol [LDL-C]) will be measured as a percentage of change from baseline. Lipids and lipoproteins will be measured at baseline, 4, 48, 96 (Day 4), and 168 (Day 7) hours, and Day 30 and Day 60.
Change From Baseline In PCSK9 At Day 60 | Baseline, Day 60
  Pharmacodynamic effects of inclisiran on PCSK9 will be measured as a percentage of change from baseline. PCSK9 protein levels will be measured at baseline, 4, 48, 96 (Day 4), and 168 (Day 7) hours, and Day 30 and Day 60.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Robson, PhD, Principal Investigator — Christchurch Clinical Studies Trust
Locations (2):
- New Zealand (2):
  - Auckland Clinical Studies Limited, Auckland
  - Christchurch Clinical Studies Trust, Christchurch

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wright RS, Collins MG, Stoekenbroek RM, Robson R, Wijngaard PLJ, Landmesser U, Leiter LA, Kastelein JJP, Ray KK, Kallend D. Effects of Renal Impairment on the Pharmacokinetics, Efficacy, and Safety of Inclisiran: An Analysis of the ORION-7 and ORION-1 Studies. Mayo Clin Proc. 2020 Jan;95(1):77-89. doi: 10.1016/j.mayocp.2019.08.021. Epub 2019 Oct 17. PMID 31630870